CLINICAL TRIAL: NCT07402226
Title: SSc-DIGEST Trial: Systemic Sclerosis DIet for GastrointESTinal Symptoms Randomized Controlled Trial of Low FODMAP, CDED, and NICE Diets for Gastrointestinal Symptoms in Systemic Sclerosis
Brief Title: Systemic Sclerosis DIet for GastrointESTinal Symptoms
Acronym: DIGEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Dinesh Khanna, MD, MS, Frederick G L Huetwell Professor of Rheumatology, Professor of Internal Medicine and Program Director, Internal Medicine, Medical School, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00285136
Record Dates: First submitted 2026-01-21; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Systemic Sclerosis (SSc)
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Microbiota

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the dietary counseling intervention, it will not be possible to blind dietitians and participants. Participants will be aware of general participation in dietary therapy but blinded to specific diet names. Investigators, outcome assessors, and the biostatistician will be fully blinded to allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diet 1: Restriction of fermentable carbohydrates (Experimental)
  Interventions: Behavioral: Diet 1: Restriction of fermentable carbohydrates
- Diet 2: Elimination of foods harmful to gut barrier and microbiome (Experimental)
  Interventions: Behavioral: Diet 2: Elimination of foods harmful to gut barrier and microbiome
- Diet 3: Regular meal patterns, soluble fiber, and portion control (Experimental)
  Interventions: Behavioral: Diet 3: Regular meal patterns, soluble fiber, and portion control

INTERVENTIONS:
Behavioral: Diet 1: Restriction of fermentable carbohydrates — 6 weeks guided diet under the supervision of a dietician restricting fermentable carbohydrates known to trigger GI symptoms.
  Arms: Diet 1: Restriction of fermentable carbohydrates
Behavioral: Diet 2: Elimination of foods harmful to gut barrier and microbiome — 6 weeks guided diet under the supervision of a dietician eliminating of foods harmful to gut barrier and microbiome
  Arms: Diet 2: Elimination of foods harmful to gut barrier and microbiome
Behavioral: Diet 3: Regular meal patterns, soluble fiber, and portion control — 6 weeks guided diet under the supervision of a dietician emphasizing regular meal patterns, soluble fiber, and portion control.
  Arms: Diet 3: Regular meal patterns, soluble fiber, and portion control

SUMMARY:
This research will evaluate the effect of diets on bloating/distention, assess changes in abdominal pain, and overall gastrointestinal symptom burden in Systemic Sclerosis. The researchers will do this by comparing outcomes of people assigned to 3 different diets. Following the research specifics of the diets will be available upon contact with the details listed below.

DETAILED DESCRIPTION:
The rationale for keeping the diets (arms/interventions names) vague is it prevents other researchers from using these diets in their studies, minimizes expectation bias of patients (who can have preference for one diet over other) and prevents participants from trying other diets before end of study period in case they don't respond.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of systemic sclerosis (SSc) as per ACR/EULAR classification criteria.• Self-reported moderate to severe gastrointestinal bloating or distension, with a UCLA SCTC-GIT 2.0 bloating Scale score ≥2.00 on (0.00-3.00 scale) at screening.
* Willingness and ability to comply with dietary intervention and study procedures.
* Ability to provide informed consent.

Exclusion Criteria:

* Diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis) or celiac disease.
* Use of systemic antibiotics within 4 weeks prior to baseline.
* History of gastrointestinal surgery (other than cholecystectomy or appendectomy unless in the last 3 months).
* Severe cognitive impairment or psychiatric illness that would limit ability to follow dietary instructions.
* Known allergy or intolerance to major components of any of the study diets (e.g., lactose, gluten) unless manageable within diet framework.
* Current or recent (within 3 months) dietary intervention for managing GI symptoms (e.g. gluten-free diet, low FODMAP diet, etc.).
* Clinically significant self-reported (≥10 percent weight loss) in the last 3 months
* BMI less than 20
* Ongoing tube feeds or TPN
* Participating in another interventional trial
* Pregnancy or lactation, or planning pregnancy in the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in Bloating severity | Baseline to week 6
  As assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.1 - Gastrointestinal Gas and Bloating 13a - 13 questions with raw summed scores ranging from 13-36.

SECONDARY OUTCOMES:
Change in Bloating severity | Baseline to week 6
  As assessed by the UCLA Scleroderma Clinical Trial Consortium Gastrointestinal Tract (UCLA SCTC GIT 2.0). The bloating score is a subsection of 4 questions with 4 options each. The score ranges from .0-3 where higher numbers indicate more frequent bloating.
Change in Abdominal pain severity | Baseline to week 6
  As assessed by the PROMIS Scale v1.0 - Gastrointestinal Belly Pain 5a - 5 questions with raw summed score range of 6-25.
Change in Overall GI symptom | Baseline to week 6
  UCLA SCTC GIT 2.0 total score (all sections but constipation) with a range of (0-2.83). Higher scores indicate more severe symtoms.

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No